CLINICAL TRIAL: NCT02012634
Title: A Multi-center, III Phase，Randomized Controlled Clinical Study of Capecitabine Metronomic Chemotherapy After Standard Adjuvant Chemotherapy in Operable Triple Negative Breast Cancer
Brief Title: Metronomic Chemotherapy of Capecitabine After Standard Adjuvant Chemotherapy in Operable Triple Negative Breast Cancer
Acronym: MACRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, LiNanlin,Ph.D, Chief Physician,Clinical Professor, The department of Vascular endocrine surgery, Xijing Hospital
Other Study IDs: TPYS-01
Record Dates: First submitted 2013-11-26; First posted 2013-12-16 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Breast Cancer; Capecitabine; Triple Negative Breast Cancer
Keywords: Breast Cancer; Capecitabine; Triple Negative Breast CancerTNBC（TNBC）
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 ml blood sample is taken before randomization
Oversight: Data Monitoring Committee: No

SUMMARY:
A Multi-center, III Phase,Randomized Controlled Clinical Study of Capecitabine Metronomic Chemotherapy After Standard Adjuvant Chemotherapy in Operable Triple Negative Breast Cancer

DETAILED DESCRIPTION:
Capecitabine comes as a tablet to take by mouth. It is usually taken twice a day (in the morning and in the evening) for 2 weeks, followed by a 1 week break before repeating the next dosage cycle. In this study, capecitabine will be prescribed as dosage of 900mg/m2, and maintain for a whole year after the standard treatment in operable triple negative breast cancer patients. DFS is set as the primary outcome, OS and DDFS are also observed as the secondary outcomes. Statistical analysis are made to see whether this metronomic therapy of capecitabine ( 900mg/m2) will bring benefit to any of the iterms above.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* aged 18 - 70 years old;
* Histological confirmed with unilateral invasive carcinoma (all pathological types are applicable);
* Newly diagnosed conditions allowing direct surgery without any absolute contraindication for surgery;
* No mass or microscopic tumor residue after surgery resection;
* Initiate adjuvant chemotherapy within 30 days after surgery;
* Axillary lymph node positive (including the sentinel lymph node positive and lymph node positive after axillary dissection), for example, axillary lymph node negative requires that primary tumor size must be greater than 1cm;
* Definite reports on ER/PR(progesterone receptor)/Her2 receptor showing all ER/PR/Her2 negative (specific definitions: immunohistochemical detection of ER <10% tumor cells is defined as ER negative, PR <10% positive tumor cells is defined as PR-negative, Her2 is 0~1+ or 2+ but determined negative via FISH or CISH detected (no amplification) is defined as Her2 negative);
* No relevant clinical or imaging evidence of metastasis showing in the preoperative examination (M0);
* Without peripheral neuropathy;
* ECOG performance score is 0 or 1;
* Postoperative recovery was good and an interval of at least one week since the surgery is necessary;
* White blood cell count> 4 × 10^9/l, neutrophil count> 2 × 10^9/l, platelet count> 100 × 10^9/l and hemoglobin 9g/dl);
* ASAT and ALAT <1.5 folds of the upper limit of normal values, alkaline phosphatase <2.5 folds of the upper limit of normal values, total bilirubin <1.5 folds of the upper limit of normal values;
* Serum creatinine <1.5 folds of the upper limit of normal value;
* Women at childbearing age should take contraception measures during treatment;
* Cardiac function: echocardiographic examination showed LEVF> 50%;
* Informed consent form signed.

Exclusion Criteria:

* Bilateral breast cancer or carcinoma in situ (DCIS / LCIS);
* Metastasis at any location;
* Any tumor > T4a (UICC1987) (accompanied by skin involvement, lump adhesion and fixation, inflammatory breast cancer);
* Any of ER, PR or Her-2 is positive;
* Contralateral breast clinically or radiologically suspected to be malignant but not confirmed which needs a biopsy;
* Previous neoadjuvant therapy, including chemotherapy, radiotherapy and hormone therapy;
* Previously suffering from malignant tumors (except for basal cell carcinoma and cervical carcinoma in situ), including contralateral breast cancer;
* Already enrolled into other clinical trials;
* Severe systemic disease and/or uncontrollable infection, unable to be enrolled in this study LEVF <50% (echocardiography);
* Suffering from severe cardiovascular and cerebrovascular diseases within six months before the randomization (such as: unstable angina, chronic heart failure, uncontrollable high blood pressure > 150/90mmHg, myocardial infarction or brain vascular accident);
* Known allergic to taxane and anthracycline agents;
* Women at childbearing age refuse to take contraception measures during the treatment and 8 weeks after completion of treatment;
* Pregnant and breast-feeding women;
* Pregnancy test showed positive results before drug administration after enrolling in to the study; With mental illness and cognitive impairment, unable to understand trial protocol and side effects and complete trial protocol and follow-ups (systematic evaluation is required before recruiting into this study);
* Without personal freedom and independent civil capacity.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients of vascular endocrine surgery department in Xijing Hospital
Sampling Method: Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
PFS（Progression-free survival） | Progression-free survival：time from the date of randomization until the date of disease progression，assessed up to 3 years
  PFS was defined as the time from the date of randomization until the date of disease progression at any site including distant metastasis or second primary tumors or death， assessed up to 3 years

SECONDARY OUTCOMES:
OS | time from the date of randomization until the date of any death occurred
  OS was defined as the time from the date of randomization until the date of any death occurred
DDFS | time from the date of randomization until the date of any disease occurred

CONTACTS AND LOCATIONS:
Overall Officials: Nanlin Li, Doctor, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital ，Fourth Military Medical University, Xi'an, Shaanxi, China